CLINICAL TRIAL: NCT02382159
Title: Observational, Retrospective, Multi-center Study for Therapeutic Practice Pattern of Lipid-lowering Drug and Its Effect on Parameters in Dyslipidemia of Type 2 Diabetes.
Brief Title: A Observational Study to Evaluate Lipid-lowering Drug Its Effect on Parameters in Dyslipidemia of Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: YYP-OS-001
Record Dates: First submitted 2015-02-25; First posted 2015-03-06 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Complex Dyslipidemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. Target disease: Patients with combined dyslipidemia accompanied by type 2 diabetes who has done exogenous visit or hospitalization from Jan 2010 to June 2014.
2. Study objective:

   1. The objective of this study is to Identifying the lipid parameter variation when treating patients who have dyslipidemia of type 2 diabetes for 3±1 months.
   2. After treating patients who have dyslipidemia of type 2 diabetes for 3±1 months, identifying the reason why changing method of drug dosage and pharmacotherapy.
   3. If the drug dosage and pharmacotherapy have been changed, Identifying the lipid parameter variation when treating patients by altered drugs for 3±1 months,

ELIGIBILITY:
Inclusion Criteria:

Among the patients, who has been hospitalized or visited the Outpatient Department OPD, who has dyslipidemia of type 2 diabetes.

1. Patients have the result of lipid parameter test at baseline and after lipid-lowering drug for at least 3 months.
2. Patients who have the result of lipid paraneter test (LDL-C ≥100mg/dL, TG ≥150mg/dL) at baseline.
3. Patients who have no received lipid lowering drug fr at least 2 months prior to the baseline.
4. Patients' age were > 20 years and <75 year.

Exclusion Criteria:

1. Patients who ahs HbA1c≥9%
2. Patients who have no the result of lipid parameter test at baseline and at baseline and after lipid-lowering drug for at least 3 months
3. Patients who have history of drug discontinuation by incresed liver enzyme or rhabdomyolysis.
4. Patients received lipid-lowering drug and TZD(Thiazolidinediones) in study period
5. Renal abnormality
6. Alcoholism or Alcohol abuse
7. Patients treated by Steroids.
8. Pregnant or lactating woman
9. Patients who are judged as not suitable for this study by Investigator.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Base-line (The starting time of treating lipid-lowering drug within 3 months period of 2010 ~ 2013 years)
     * Background of Patients: Basic information(Height, Weight), Smoking, Drinking and other related illness.
     * Hypoglucemic agent, Diabetes test(Fasting blood glucose, GL test, Glycated Hemoglobin)
     * At the time of Starting the treating lipid-lowering drug, total Cholesterol, TG, LDL-C, HDL-C checked before treating lipid-lowering drug.
  2. After 3±1 months from base-line
     * Hypoglycemic agent, Diabetes test
     * Total Cholesterol, TG, LDL-C at the point of 3±1 months from treating changed lipid-lowering drug, and the reason of drug dosage and pharmacotherapy
  3. After 3±1 months from treating by changed lipid-lowering drug
     * Hypoglycemic agent, Diabetes test
     * Total Cholesterol, TG, LDL-C, HDL-C at the point of 3±1 months from treating changed lipid-lowering drug.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Variation of the Lipid parameter pattern patients who are treated by lipid-lowering drug. | Over 3±1 months
  Increasing LDL-C + Triglyceride(TG)Decreasing HDL-C + Increasing TG

SECONDARY OUTCOMES:
The reason why changed drug dosage and pharmacotherapy after patients taken lipid-lowering drug. | Over 3±1 months
  Increasing LDL-C + TG Decreasing HDL-C + Increasing TG
Variation for lipid parameter when the patients who are treated for 3±1 months by lipid-lowering drug. | Over 3±1 months
  Increasing LDL-C + TGDecreasing HDL-C + Increasing TG

OTHER OUTCOMES:
Setting the sub-group by the result of lipid parameter | Basis on the Base-line
  Decreasing HDL-C: HDL-C≤40mg/dL(Man), ≤50mg/dL(Woman) Non-decreasing HDL-C: HDL-C≤40mg/dL(Man), >50mg/dL(Woman)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Rae Kim, M.D, Principal Investigator — Catholic University of Korea (Bucheon St.Mary's Hospital)
Locations (1):
- The Catholic University of Korea(Bucheon St. Mary's Hospital), Bucheon-si, South Korea